CLINICAL TRIAL: NCT06593288
Title: Randomized Clinical Trial of Spontaneous Breathing Test
Brief Title: Trial of Spontaneous Breathing Test
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ana Carlotti, Faculty of Medicine of Ribeirao Preto, University of Sao Paulo, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 82637424.6.1001.5440
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Mechanical Ventilation; Spontaneous Breathing Trial; Extubation Readiness; Extubation Failures; Pediatrics
Keywords: spontaneous breathing trial; extubation readiness test; mechanical ventilation; pediatric intensive care
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with 2 arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spontaneous breathing trial with pressure support (Active Comparator): Spontaneous breathing trial with pressure support
  Interventions: Other: Pressure Support Ventilation
- Spontaneous breathing trial without pressure support (Active Comparator): Spontaneous breathing trial without pressure support ( CPAP)
  Interventions: Other: continuous positive airway pressure (CPAP)

INTERVENTIONS:
Other: Pressure Support Ventilation — Conduct the Spontaneous breathing trial with pressure support
  Arms: Spontaneous breathing trial with pressure support
Other: continuous positive airway pressure (CPAP) — Conduct the spontaneous breathing trial with CPAP
  Arms: Spontaneous breathing trial without pressure support

SUMMARY:
The hypothesis is that the Spontaneous Breathing Test (SBT) without pressure support (PS) is not inferior to the SBT with pressure support in relation to the following outcomes: a) extubation failure; b) time on MV.

The main objective of this study is to determine whether SBT without PS is non-inferior to SBT with PS in relation to the primary outcome: a) extubation failure; and secondary outcomes: b) length of stay in the PICU and c) days free of MV.

Pacients will be randomized to 2 arms:

1. SBT with PS
2. SBT without PS (with PEEP only)

DETAILED DESCRIPTION:
Introduction Mechanical ventilation (MV) is a common procedure for patients admitted to pediatric intensive care units (PICUs). Although MV is often necessary and life-saving, it can be associated with complications such as ventilator-associated pneumonia, cardiovascular dysfunction, airway injury, and patient immobility. The longer the duration of MV, the greater the risk of morbidity, length of stay, and mortality. To reduce the risks associated with prolonged MV, clinicians should seek to continually optimize the process of weaning from ventilation (WVL), thereby increasing the likelihood of successful extubation. WVL is defined as "the gradual reduction of mechanical ventilatory support and the transfer of respiratory control and the work of breathing back to the patient." Traditionally, WVL was conducted through clinical judgment and a personal decision. Only in recent years have protocol-based approaches been implemented, with conflicting results, although most studies show that a protocolized approach tends to reduce the duration of mechanical ventilation. Extubation is defined as "removal of the endotracheal tube," and extubation failure occurs when a patient requires reintubation within hours or days of a planned extubation. More recently, extubation failure has been considered as reintubation within 48 hours of a planned extubation. Extubation failure may be secondary to the inability to maintain alveolar oxygenation and/or ventilation, airway patency and protection, secretion control, or any combination of these. Extubation failure occurs in 3-22% of patients regardless of the severity of the underlying disease, with evidence that its occurrence can directly worsen patient outcomes, including an increased mortality rate. Various clinical approaches are used to decide the best timing for extubation, ranging from the use of tools such as chest and diaphragm ultrasound to readiness testing and spontaneous breathing, but there is no clear evidence on which technique is best in children.

Rationale

When using MV, it is important to critically balance the minimization of procedural risks against the risks of extubation failure (EF) and its association with morbidities. The International Guidelines for Liberation from Mechanical Ventilation in Pediatrics were published in 2022 with the aim of guiding best practices for liberation from MV.(2) Experts have given their opinions on the various aspects of liberation from MV. Among several definitions, the most important for this study are:

Extubation readiness test (ERT): (95.7% agreement). It is a set of elements (bundle) that are used to assess the patient's eligibility to be liberated from invasive MV (IMV). In addition to the usual ERT components, such as values of the fraction of inspired oxygen (FiO2), positive end-expiratory pressure (PEEP), the factor that led to tracheal intubation in resolution, ERT may include factors such as: assessment of the level of sedation; neurological adequacy of airway control (coughing and choking); probability of upper airway obstruction after extubation; assessment of respiratory muscle strength; magnitude of airway secretions; hemodynamic status and planning of respiratory support after extubation Spontaneous breathing trial (SBT): (91.3% agreement). Systematic method of reducing IMV support to predetermined parameters to assess the likelihood that the patient will be able to independently maintain minute ventilation and gas exchange without excessive respiratory effort, if released from IMV.

Among the recommendations of the guidelines:

* Recommendation 1. A protocolized assessment was suggested to assess eligibility for SBT (100% agreement). - Notes: SBT should be conducted at regular intervals to identify when the patient has met pre-established parameters to conduct safe extubation.
* Recommendation 2. The protocolized use of the SBT bundle was suggested compared to the clinical assessment of readiness for extubation (88% agreement). - Notes: The EBT bundle includes elements that are used to assess whether the patient is ready to be released from IMV. In addition to the SBT, it may include factors such as assessment of sedation, adequacy of neurological control of the airway (coughing and choking), likelihood of upper airway obstruction, assessment of respiratory muscle strength, magnitude of airway secretions, hemodynamic status, and planning of respiratory support after extubation.
* Recommendation 3. It was suggested that the SBT be performed as part of the EBT bundle to objectively assess whether the patient is able to independently maintain adequate minute ventilation and gas exchange without excessive respiratory effort if released from IMV (96% agreement).
* Recommendation 4. It was suggested that pressure support (PS) be increased with CPAP or CPAP alone during the SBT in mechanically ventilated children at standard risk of extubation failure (Conditional recommendation, with very low level of evidence).
* Recommendation 5. For children at high risk of extubation failure (Table 1), it was suggested to use CPAP without increasing PS during SBT to better assess readiness for extubation (Conditional recommendation, with very low level of evidence).

Since the levels of evidence are low on how to perform SBT (with or without PS), there is a knowledge gap. In clinical practice, studies show the use of SBT with PS by most clinicians. Khemani et al. advocate that SBT should be performed without pressure support. Ferguson et al. in a study of 755 extubations concluded that an SBT using pressure support set at higher levels for smaller endotracheal tubes overestimates readiness for extubation in children and contributes to a higher rate of unsuccessful extubation.

Hypothesis The hypothesis is that the Spontaneous Breathing Trial without pressure support is not inferior to the Spontaneous Breathing Trial with pressure support in relation to the following outcomes: a) extubation failure; b) time on MV.

General Objective The main objective of this study is to determine whether the SBT without PS is not inferior to the SBT with PS in relation to the primary outcome: a) extubation failure; and secondary outcomes: b) length of stay in the PICU and c) days free of MV (DLMV).

Study Design/Methodology The study will be multicenter, randomized, open-label, prospective, with two arms. The study will be submitted to the Research Ethics Committee of all centers and authorization will be requested from the patients' parents or legal guardians by signing the informed consent form (ICF). The study will be registered on Clinicaltrials.gov and will follow the CONSORT 2010 guidelines. Patients admitted to participating PICUs receiving IMV for more than 24 hours will be screened twice a day (between 7:00 and 9:00 a.m.; between 2:00 and 4:00 p.m. in the afternoon) for the Extubation Readiness Test (EBT) and, if they pass, will proceed to the Spontaneous Breathing Trial (SBT) lasting one hour.

Inclusion criteria:

* Patients admitted to the PICU on IMV for more than 24 hours
* Patients over 1 month of age (corrected gestational age > 38 weeks) and < 18 years old on the day of screening for ERT

Exclusion criteria:

* Perinatal-related lung disease
* Congenital diaphragmatic hernia or congenital/acquired paralysis of the diaphragm
* Children with heart disease
* Primary pulmonary hypertension
* Bronchiolitis obliterans
* Post-hematopoietic stem cell transplant; specifically, patients receiving continuous supplemental oxygen for three or more days prior to intubation; receiving noninvasive ventilation for more than 24 hours prior to intubation; receiving more than one vasoactive medication at the time of meeting the inclusion criteria; spending more than four days in the PICU prior to intubation; supported on or with immediate plans for renal replacement therapies; with two or more allogeneic transplants; who relapsed after transplant; or with diffuse alveolar hemorrhage
* Post-lung transplantation
* Home ventilator dependence with baseline Oxygen Saturation Index (OSI) >6 (baseline is defined as a stable period prior to the present illness)
* Neuromuscular respiratory failure
* Critical airway obstruction (e.g., post-laryngotracheal surgery or new tracheostomy) or anatomical lower airway obstruction (e.g., mediastinal mass)
* Facial surgery or trauma in the past two weeks
* Intracranial bleeding
* Morbid obesity (2w-24mo: WHO weight-for-length z-score/height z-score ≥+3; ≥2y: WHO body mass index (BMI)-for-age z-score ≥+3)
* Family/medical team unsupportive total (patient treatment considered futile)
* Previously enrolled in a current study
* Enrolled in any other clinical trial with intervention not approved for concomitant enrollment
* Pregnancy

Extubation Readiness Test: This is a standardized test to determine whether the patient is ready to be extubated from a pulmonary perspective. The test should not be initiated if:

* There is no neurological responsiveness and the ability to protect the airway is altered
* Inaudible air leak around an uncuffed/deflated COT
* Scheduled procedure requiring deep sedation/anesthesia (e.g., MRI, surgery, etc.)

Patients who meet the following prerequisites will be considered eligible for extubation:

* Spontaneous breathing
* IO/ISO ≤ 6
* Reduction and/or stabilization of ventilator support in the last 12 hours

In this case, proceed to the checklist (yes/no):

* Cause of intubation in resolution
* Cardiovascular stability/vasoactive drugs in reduction/discontinued
* May have altered creatinine, but must be urinating/without fluid overload. - No excess secretions (22)
* No change in level of consciousness and no respiratory effort
* MV parameters: FIO2≤50% PEEP≤8 PIP≤25 If all the above requirements are met, the patient will be able to undergo SBT.* *SBT may be postponed by the attending physician, even if all prerequisites are met, if he/she believes that the patient is not clinically well or has an upcoming procedure to be performed while intubated (e.g., Magnetic Resonance Imaging)

Patients who passed the TPE and are able to undergo SBT will be randomized to:

Arm 1: SBT (1 hour) with PEEP and without PS. The patient should remain with the same PEEP and FiO2 as during the TPE.

Arm 2: SBT (1 hour) with PEEP and with PS. The patient should remain with the same PEEP and FiO2 as during the TPE. The PS will be adjusted according to the diameter of the tracheal tube.

PS= 6cmH2O for TOT > 5mm PS= 8cmH2O for TOT 4 - 5mm PS= 10cmH2O for TOT ≤ 3.5mm

The following parameters must be monitored and recorded on a form (Appendix I): HR, RR, SatO2, respiratory effort at times zero, five, ten, twenty, thirty, forty-five and sixty minutes.

The SBT will be considered failed if:

* There is a drop in SatO2 <92% maintained for 5 minutes;
* Increase in RR maintained for 5 minutes above normal for age;
* Increase in HR maintained for 5 minutes above normal for age;
* Increase in respiratory effort maintained for 5 minutes (consensus between physiotherapist and attending physician); Otherwise, the SBT will be considered positive and the patient must progress to tracheal extubation.

If the patient passes the SBT and does not progress to tracheal extubation, the reason must be stated on the study form.

After tracheal extubation

* May extubate to a higher FiO2 than on the ventilator and then reduce FiO2 every 2 hours to maintain SpO2≥94%
* If the patient develops respiratory distress after extubation:

  * If stridor is present: consider IV dexamethasone + epinephrine inhalation Q15 min
  * If stridor is not present: consider NIV or LEEP

Extubation failure Early extubation failure will be defined as the participant being reintubated within 48 hours after the planned tracheal extubation.

Randomization When patients meet the study inclusion criteria, the informed consent form will be applied to parents/guardians.

Once the informed consent form has been signed, randomization will be carried out using the REDCap tool.

Statistical Analysis Descriptive data will be expressed as frequencies (%). The distribution of each continuous variable will be described by medians and interquartile ranges (IQRs). The Mann-Whitney U test and the Chi-Square test or Fisher's exact test will be used to compare continuous and nominal variables, respectively. The Kruskal-Wallis test will be used to compare continuous variables between more than two groups.

Sample size calculation

The null hypothesis to be tested is that the percentage of successful extubation for patients on pressure support is better than the percentage for those on CPAP, above a tolerance value of 10% or 15% (delta, or non-inferiority limit):

H0: πps ≥ πcpap + d, where πs = percentage of successful extubation on pressure support; πcpap = percentage of successful extubation on CPAP; d = delta tolerance (10% or 15%). By rejecting H0, the alternative hypothesis is accepted that the percentage for those on CPAP is πs - d : H1 : πps - d < πcpap.

Therefore, by accepting H1, it is confirmed that CPAP is not inferior to pressure support, within the margin of tolerance.

In the study by Ferguson et al., 755 extubation readiness tests were performed on 538 patients using pressure support. 5.8% required reintubation (success rate of 94.2%).(16) Using the success rates from this study for our sample size calculation, 94 patients will be needed in each group (188 patients for both arms) to show with 90% power (1-beta) that the upper limit of a two-sided 90% confidence interval (or 95% of a one-sided CI) will exclude a difference in favor of the Pressure Support group for a delta of 10%.

42 patients will be needed in each group (84 patients for both arms) for a delta of 15% and a power of 90%.

For a power of 80% and a delta of 10%, 68 patients will be needed in each group (136 patients for both arms). For a power of 80% and a delta of 15%, 31 patients will be needed in each group (62 patients for both arms).

Considering an estimated loss of 20% of the sample due to various causes (medical record problems, participant withdrawals and unforeseen causes), considering a power of 80% and a delta of 10%, it is expected to recruit 170 patients in both arms of the study.

To determine non-inferiority, it will be used the Farrington-Manning test from the DescrTab2 package of R: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna.

Study Location A multicenter study, with the Hospital das Clínicas of the Ribeirão Preto Medical School of the University of São Paulo (FMRP-USP) as the proposing institution. The other participating centers will be invited to join the study through an invitation made by the Brazilian Research Network in Pediatric Intensive Care (Brnet-PIC) to reach the required sample size.

Ethical Issues A free and informed consent form (FICF) will be applied to the research participants, signed by a parent or guardian during the study. For participants over 6 years of age, the free and informed consent form (FICF) will also be applied, which may be applied later, since the patients will be sedated and on MV during randomization.

Risks and benefits Risks: although unlikely, there may be risks related to the breach of data confidentiality. However, the researchers will undertake to take all possible measures to maintain the confidentiality of the data of the study subjects. Confidentiality will be maintained by the anonymity of the questionnaire and by the division of hospitals by region of the country and not by their name or specific geographic location. In principle, choosing a support mode in a given arm of the study over the other arm does not imply any risk to the patient.

Benefits: the results of this study will not bring a direct benefit to the study participants, but may bring benefits in expanding knowledge regarding best practices for safe extubation of future patients.

Data Management and Protection Data will be collected through electronic forms from REDCap (Research Electronic Data Capture, Vanderbilt, USA) and participants will have their data de-identified. Data storage will be handled by the University of São Paulo and protected by an encrypted password. Digital forms will be deleted from any data source after a regulatory period of five years.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the PICU on MV for more than 24 hours
* Patients over 1 month old (corrected gestational age > 38 weeks) and < 18 years old on the day of screening for ERT

Exclusion Criteria:

* Perinatal-related lung disease
* Congenital diaphragmatic hernia or congenital/acquired paralysis of the diaphragm
* Children with heart disease
* Primary pulmonary hypertension
* Bronchiolitis obliterans
* Post-hematopoietic stem cell transplant; specifically, patients receiving continuous supplemental oxygen for three or more days prior to intubation; receiving noninvasive ventilation for more than 24 hours prior to intubation; receiving more than one vasoactive medication at the time of meeting the inclusion criteria; spending more than four days in the PICU prior to intubation; supported by or with immediate plans for renal replacement therapy; with two or more allogeneic transplants; who relapsed after transplant; or with diffuse alveolar hemorrhage
* Post-lung transplantation
* Home ventilator dependence with baseline Oxygen Saturation Index (OSI) >6 (baseline is defined as a stable period prior to the present illness)
* Neuromuscular respiratory failure
* Critical airway obstruction (e.g., post-laryngotracheal surgery or new tracheostomy) or anatomical lower airway obstruction (e.g., mediastinal mass)
* Facial surgery or trauma in the past two weeks
* Intracranial bleeding
* Morbid obesity (2w-24mo: WHO weight-for-length z-score/height z-score ≥+3; ≥2y: WHO body mass index (BMI)-for-age z-score ≥+3)
* Family/medical team unsupportive total (patient treatment considered futile)
* Previously enrolled in a current study
* Enrolled in any other clinical trial with intervention not approved for concomitant enrollment
* Pregnancy

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Extubation failure | 48 hours
  Extubation failure: patient needs to be reintubated less than 48 hours after extubation

SECONDARY OUTCOMES:
Free days of mechanical ventilation | 30 days
  Free days of mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Ana Paula C Carlotti, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto da Universidade de Sao Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Brazil's law prohibits sharing participants data

REFERENCES:
- [Derived] Colleti Junior J, Araujo OR, Weber KT, Santos GMVD, Silva DCBD, Volpon LC, Carlotti APCP. Protocol for a non-inferiority randomized controlled trial of spontaneous breathing trial in children with and without pressure support. Crit Care Sci. 2025 Dec 15;37:e20250187. doi: 10.62675/2965-2774.20250187. eCollection 2025. PMID 41417398